CLINICAL TRIAL: NCT03774537
Title: Intravenous Human Umbilical-Cord-Derived Mesenchymal Stem Cells For Premature Infants Ａt High Risk For Bronchopulmonary
Brief Title: Human Mesenchymal Stem Cells For Infants At High Risk For Bronchopulmonary Dysplasia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xia Yunqiu, Director, Children's Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XiaYQ
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: high risk； Bronchopulmonary Dysplasia；hUC-MSCs
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transplantation of hUC-MSCs (Experimental): Preterm infants at high risk for BPD will receive transplantation of hUC-MSCs.
  Interventions: Drug: Transplantation of hUC-MSCs
- No transplantation of hUC-MSCs (Other): Preterm infants at high risk for BPD will not receive transplantation of hUC-MSCs
  Interventions: Drug: No transplantation of hUC-MSCs

INTERVENTIONS:
Drug: Transplantation of hUC-MSCs — Preterm infants at high risk for BPD will receive transplantation of hUC-MSCs through intravenous infusion. Dose A - 1 million cells per kg; Dose B - 5 million cells per kg
  Other Names: Intravenous infusion of hUC-MSCs
  Arms: Transplantation of hUC-MSCs
Drug: No transplantation of hUC-MSCs — Preterm infants at high risk for BPD will not receive transplantation of hUC-MSCs
  Other Names: No intravenous infusion of hUC-MSCs
  Arms: No transplantation of hUC-MSCs

SUMMARY:
This study is an open-label, single-center, dose escalation study to evaluate of safety and efficacy of human umbilical cord -derived mesenchymal stem cells (hUC-MSCs) in premature infants at high risk for Bronchopulmonary Dysplasia（BPD）

DETAILED DESCRIPTION:
BPD is a chronic lung disease that occur in premature infants receiving prolonged oxygen pulmonary and ventilator therapy. It remains a main complication of extreme prematurity and currently lacks efficient treatment.The mortality rate of one year after birth is still high and the quality of life is not optimistic.

hUC-MSCs are widely used in clinic due to their low immunogenicity and convenient to get. Many animal study had shown that hUC-MSCs had therapeutic effects on a variety of animal models of lung disease.Furthermore,there are a large number of clinical trials of MSCs applied to various system diseases and the safety was verified.So, the main purpose of this study is to evaluate the safety and efficacy of hUC-MSCs in participants at high risk for BPD

ELIGIBILITY:
Inclusion Criteria:

1. An infant whose postnatal age is 3 to 14 days, inclusive (for treatment between 5 and 14 days after birth)
2. Gestational age is between 23 and 28 weeks (23 weeks ≤ gestational age (GA) < 28 weeks)
3. Birth weight is between 500g and 1000g, inclusive
4. Being intubated and receiving mechanical ventilation within 5-14 days after birth, with a fraction of inspired oxygen (FiO2) of 0.25 or greater at Screening
5. Written consent form signed by a legal representative or a parent.

Exclusion Criteria:

1. Although mechanical ventilation or oxygen is required in participants, there are no signs of dyspnea or BPD-related changes in lung imaging, such as central apnea or diaphragm paralysis.
2. The participants who have complex congenital heart disease.
3. The participants who have severe pulmonary hypertension(cardiac ultrasound confirmed) at the time of assessment.
4. The participants who have severe respiratory tract malformation: pierre-robin syndrome, tracheobronchomalacia, vascular ring syndrome, congenital tracheal stenosis, tracheo-esophageal fistula, pulmonary emphysema, pulmonary sequestration, congenital pulmonary dysplasia, congenital pulmonary cyst, congenital spasm, etc.
5. The participants who have severe chromosome anomalies :Edward syndrome, Patau syndrome, Down syndrome, etc) or severe congenital malformation (Hydrocephalus, Encephalocele, etc).
6. The participants who have severe congenital infection(Herpes, Toxoplasmosis, Rubella, Syphilis, AIDS, etc).
7. The participants who have severe sepsis or shock.
8. The participants who is going to have surgery 72 hours before/after this study drug administration.
9. The participants who have surfactant administration within 24 hours before this study drug administration.
10. The participants who have severe intracranial hemorrhage ≥ grade 3 or 4.
11. The participants who have active pulmonary hemorrhage or active air leak syndrome at the time of assessment.
12. The participants who have the history of other clinical studies as a participant.
13. The participants who is considered inappropriate by the investigators.

Ages: 4 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse reactions related to infusion after treatment | 24 hours after administration
  To evaluate the safety of hUC-MSCs for BPD.

SECONDARY OUTCOMES:
The incidence and severity of BPD defined by the National Institutes of Child Health and Human Development (NICHD) workshop. | at the corrected gestational age of 36 weeks
  To evaluate the efficacy of hUC-MSCs to prevent preterm infants at high risk of BPD from developing BPD
Changes of high-resolution chest CT in participants | within 2 years after administration
  To evaluate the safety and efficacy of human umbilical cord -derived mesenchymal stem cells for BPDmesenchymal stem cells for BPD.
Changes of temperature in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD.mesenchymal stem cells for BPD.
Changes of blood pressure in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD. Blood pressure is measured by electronic sphygmomanometer.
Changes of respiratory rate in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD.
Changes of oxygen saturation in participants | 3 days after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for BPD.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Fu, Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang YS, Ahn SY, Yoo HS, Sung SI, Choi SJ, Oh WI, Park WS. Mesenchymal stem cells for bronchopulmonary dysplasia: phase 1 dose-escalation clinical trial. J Pediatr. 2014 May;164(5):966-972.e6. doi: 10.1016/j.jpeds.2013.12.011. Epub 2014 Feb 6. PMID 24508444
- [Background] Hayes D Jr, Meadows JT Jr, Murphy BS, Feola DJ, Shook LA, Ballard HO. Pulmonary function outcomes in bronchopulmonary dysplasia through childhood and into adulthood: implications for primary care. Prim Care Respir J. 2011 Jun;20(2):128-33. doi: 10.4104/pcrj.2011.00002. PMID 21336467
- [Background] Ahn SY, Chang YS, Kim JH, Sung SI, Park WS. Two-Year Follow-Up Outcomes of Premature Infants Enrolled in the Phase I Trial of Mesenchymal Stem Cells Transplantation for Bronchopulmonary Dysplasia. J Pediatr. 2017 Jun;185:49-54.e2. doi: 10.1016/j.jpeds.2017.02.061. Epub 2017 Mar 21. PMID 28341525
- [Background] Wilson JG, Liu KD, Zhuo H, Caballero L, McMillan M, Fang X, Cosgrove K, Vojnik R, Calfee CS, Lee JW, Rogers AJ, Levitt J, Wiener-Kronish J, Bajwa EK, Leavitt A, McKenna D, Thompson BT, Matthay MA. Mesenchymal stem (stromal) cells for treatment of ARDS: a phase 1 clinical trial. Lancet Respir Med. 2015 Jan;3(1):24-32. doi: 10.1016/S2213-2600(14)70291-7. Epub 2014 Dec 17. PMID 25529339
- [Background] Laube M, Stolzing A, Thome UH, Fabian C. Therapeutic potential of mesenchymal stem cells for pulmonary complications associated with preterm birth. Int J Biochem Cell Biol. 2016 May;74:18-32. doi: 10.1016/j.biocel.2016.02.023. Epub 2016 Feb 27. PMID 26928452
- [Background] Pierro M, Ionescu L, Montemurro T, Vadivel A, Weissmann G, Oudit G, Emery D, Bodiga S, Eaton F, Peault B, Mosca F, Lazzari L, Thebaud B. Short-term, long-term and paracrine effect of human umbilical cord-derived stem cells in lung injury prevention and repair in experimental bronchopulmonary dysplasia. Thorax. 2013 May;68(5):475-84. doi: 10.1136/thoraxjnl-2012-202323. Epub 2012 Dec 4. PMID 23212278
- [Background] Hansmann G, Fernandez-Gonzalez A, Aslam M, Vitali SH, Martin T, Mitsialis SA, Kourembanas S. Mesenchymal stem cell-mediated reversal of bronchopulmonary dysplasia and associated pulmonary hypertension. Pulm Circ. 2012 Apr-Jun;2(2):170-81. doi: 10.4103/2045-8932.97603. PMID 22837858
- [Background] Yeh TF, Chen CM, Wu SY, Husan Z, Li TC, Hsieh WS, Tsai CH, Lin HC. Intratracheal Administration of Budesonide/Surfactant to Prevent Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2016 Jan 1;193(1):86-95. doi: 10.1164/rccm.201505-0861OC. PMID 26351971